CLINICAL TRIAL: NCT05928715
Title: Effect of Finger Feeding on Term Newborns: A Randomized Controlled Study
Brief Title: Effect of Finger Feeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Amasya University (Other)
Collaborators: Mustela Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 106728
Record Dates: First submitted 2023-03-30; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-03

CONDITIONS: Finger Feeding; Alternative Feeding Methods
Keywords: Finger Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): It is the group that will receive breast milk or formula by finger feeding.
  Interventions: Other: Finger feeding
- Control group (No Intervention): No Intervention: control group attempt will not be implemented

INTERVENTIONS:
Other: Finger feeding — The newborn will receive every expressed breast milk or formula support during the day with the finger feeding method.
  Arms: Experimental group

SUMMARY:
With the planned study, it was aimed to determine the effect of finger feeding method on newborns in term babies.

DETAILED DESCRIPTION:
It was planned as a randomized controlled experimental study design.

Full randomization will be performed and infants who meet the inclusion criteria will be assigned to groups by flipping a coin.

On the toss of a coin, if heads came up then subject was allocated to the control group. If tails came up, then subject was allocated to the intervention group. This procedure was repeated for each mother.

Within the scope of the study, "Informed consent" will be obtained from the parents for infants who need formula supplementation or for infants fed with expressed breast milk by the decision of the Physician in the experimental and control groups.

Babies in the control group will continue to receive routine care and no intervention will be made on their feeding style. The researcher will be informed verbally and practically about the finger feeding method and the application steps to the mothers of the babies in the experimental group and to the family members who will support their feeding in baby care. In this direction, it will be ensured that expressed breast milk or formula support is given by finger feeding method.

ELIGIBILITY:
Inclusion Criteria:

Mother is 18 years or older Newborns 38 weeks and older Newborns who do not have any postnatal health problems and are followed up with the mother Babies taking formula supplements Babies who have difficulty breastfeeding There is no obstacle to breastfeeding or breastfeeding

Exclusion Criteria:

Babies with sucking and swallowing dysfunction Babies with respiratory distress (respiratory rate over 60/min, babies with groaning, nasal wing breathing)

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding | 15 days after the start of the intervention
  Number of breastfeeding per day
Expressed breast milk | 15 days after the start of the intervention
  amount of daily expressed breast milk intake
Formula intake | 15 days after the start of the intervention
  amount of daily formula consumption
finger feeding | 15 days after the start of the intervention
  number of finger feeding per day

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University Faculty of Health Sciences, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It will be shared if requested and deemed appropriate.